CLINICAL TRIAL: NCT06098781
Title: Patient Reported Outcomes After Gynaecological Gender Surgeries
Brief Title: Gynaecological Gender-affirming Surgeries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, J.A.F. Huirne, Professor, Amsterdam UMC, location VUmc
Other Study IDs: 2020.332
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Gender Dysphoria
Keywords: hysterectomy; colpectomy; vaginectomy; tubectomy; patient-reported outcome measure
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective cohort study is to learn about the patient report outcomes after gynaecological gender-affirming surgeries (i.e. hysterectomy, tubectomy, colpectomy) among trans-masculine and non-binary individuals (assigned female at birth).

The main question it aims to answer are:

• What is the experienced effect of gynaecological gender-affirming surgeries

Participants will be asked to fill out a questionaire pre-operatively and 3,9 and 18 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* assigned female at birth
* scheduled to undergo gynaecological gender-affirming surgery (i.e. hysterectomy, ovariectomy, tubectomy and/or colpectomy)

Exclusion Criteria:

* age below 18 y/o
* surgery combined with other surgeries (e.g. urethroplasty, metoidioplasty)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Trans-masculine or non-binary individuals (assigned female at birth)
Study Population: Trans-masculine or non-binary individuals (assigned female at birth) with wish to undergo gynaecological gender-affirming surgeries
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Experienced effect on gender dysphoria | 3& 9 months
  On a scale of -5 to +5 the experienced effect on gender dysphoria
Experienced effect on gender dysphoria measured by GCLS | 9 & 18 months
  Comparison of GCLS score (gender congruence life satisfaction scale) pre-operatively and post-operatively

SECONDARY OUTCOMES:
Experienced effect on psychological well being | 3 & 9 months
  On a scale of -5 to +5 the experienced effect on psychological well being
Experienced effect on confidence | 3& 9 months
  On a scale of -5 to +5 the experienced effect on confidence
Experienced effect on sexual experience | 3& 9 months
  On a scale of -5 to +5 the experienced effect on sexual experience
Surgical satisfaction | 3& 9 months
Impact of health on satisfaction of life | 3 & 9 months
  Comparison of Short Form Health Survey (SF12) pre- and postoperatively
Physical complaints post-operatively | 3 & 9 months
  physical complaints (bleeding, discharge, abdominal/pelvic pain, difficulty sitting, difficulty peeing, climacterial other complaints)
Recovery time postoperatively | 3 months
  Time to recovery of daily activities

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Location VU Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided